CLINICAL TRIAL: NCT03048513
Title: Clinical Presentation of Melioidosis in Head and Neck Region
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Principal investigator, Khon Kaen University
Other Study IDs: MEC007/59
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Melioidosis; Head and Neck Infection
Keywords: Melioidosis; Head and Neck; Clinical
MeSH Terms: conditions — Melioidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient who presented with melioidosis in head and neck — Investigators assess the patients who had the pus culture positive with Burkholderia pseudomallei.

SUMMARY:
Melioidosis in head and neck was observed including clinical presentation, diagnosis with titer, and result of treatment.

DETAILED DESCRIPTION:
This research is retrospective study about five years ( Jan 2011- Oct 2016).

ELIGIBILITY:
Inclusion Criteria:

* Patients who has the pus culture from head and neck region positive with Burkholderia pseudomallei

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who has the pus culture from head and neck region positive with Burkholderia pseudomallei. Furthermore, these pateints were received treatment at Mukdahan Hospital, Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Location of infection in head and neck as assess by clinical diagnosis | 5 years
  These results will be reported as single or multiple site infection in head and neck region.

SECONDARY OUTCOMES:
Diagnosis as confirm with pus culture | 5 years
  Assessing the correlation of melioid titer and culture by Pearson statistic
Number of participants with successful treatment as assess by clinical presentation | 5 years
  These results will be evaluated as remission or recurrent. The remission mean that fever or pus collection is subside and no presentation with melioidosis again in 5 years.
  The recurrent mean that participants will present with clinical melioidosis again in 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dance DA, Davis TM, Wattanagoon Y, Chaowagul W, Saiphan P, Looareesuwan S, Wuthiekanun V, White NJ. Acute suppurative parotitis caused by Pseudomonas pseudomallei in children. J Infect Dis. 1989 Apr;159(4):654-60. doi: 10.1093/infdis/159.4.654. PMID 2926159